CLINICAL TRIAL: NCT05761795
Title: A Randomized, Controlled, Double-Masked Adaptive Design Evaluation of the Safety and Preliminary Efficacy of IVMED-85 on Pediatric Myopia
Brief Title: Efficacy of IVMED-85 on Pediatric Myopia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: iVeena Delivery Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IVNA 22-01
Record Dates: First submitted 2023-02-23; First posted 2023-03-09 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- IVMED-85 Low Dose and placebo (Experimental): Total subjects n=6 n=4 IVMED 85 Low Dose n=2 placebo BID for 1 month
  Interventions: Drug: IVMED 85; Drug: Placebo
- IVMED-85 Mid Dose and placebo (Experimental): Total subjects n=6 n=4 IVMED 85 Mid Dose n=2 placebo BID for 1 month
  Interventions: Drug: IVMED 85; Drug: Placebo
- IVMED-85 High Dose and placebo (Experimental): Total subjects n=6 n=4 IVMED 85 High Dose n=2 placebo BID for 1 month
  Interventions: Drug: IVMED 85; Drug: Placebo
- IVMED-85 Low Dose (Experimental): Total subjects n=48 IVMED 85 Low Dose BID for 12 month
  Interventions: Drug: IVMED 85
- IVMED-85 Mid Dose (Experimental): Total subjects n=48 IVMED 85 Mid Dose BID for 12 month
  Interventions: Drug: IVMED 85
- IVMED-85 High Dose (Experimental): Total subjects n=48 IVMED 85 High Dose BID for 12 month
  Interventions: Drug: IVMED 85
- Placebo (Placebo Comparator): Total subjects n=54 Placebo BID for 12 month
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IVMED 85 — Eye drop
  Arms: IVMED-85 High Dose; IVMED-85 High Dose and placebo; IVMED-85 Low Dose; IVMED-85 Low Dose and placebo; IVMED-85 Mid Dose; IVMED-85 Mid Dose and placebo
Drug: Placebo — Placebo eye drop
  Arms: IVMED-85 High Dose and placebo; IVMED-85 Low Dose and placebo; IVMED-85 Mid Dose and placebo; Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety and preliminary efficacy of a 1-year course of IVMED-85 eye drops for the treatment of pediatric myopia by assessing its safety effects on visual acuity and its effect on the change and/or progression of myopia.

The main question[s] it aims to answer are:

* Does IVMED 85 improve visual acuity
* Does IVMED 85 slow or otherwise change the progression of myopia

Participants will use eyedrops twice a day for one year. Researchers will compare IVMED 85 to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* To be considered for enrollment in the study, the patient must meet all of the following criteria:

  1. Age 5 to 16 years and 6 months, three age groups cohorts (5-8), (9-12), and (13-16) (Phase 1 patients will be exclusively age 13-16).
  2. Refractive error by cycloplegic refraction in both eyes: myopia -0.75 D to -9.75 D spherical equivalent; astigmatism ≤ 4.00D; anisometropia <3.00 D
  3. Best corrected distance visual acuity better than or equal to Snellen 20/40 (logMAR equivalent 0.3) in both eyes
  4. Kmax >40 D and <50 D in both eyes
  5. Minimum corneal thickness > 350 microns in both eyes
  6. Absence of ocular comorbidities (glaucoma, cataract, anterior segment dysgenesis, corneal scarring, juvenile rheumatoid arthritis, lens subluxation, uveitis, collagen disorders (Ehlers-Danlos, Marfan's syndrome, osteogenesis imperfecta, retinal diseases) in both eyes
  7. Written informed consent from a parent or legal guardian and assent from participant
  8. Willing and able to comply with clinic visits and study-related procedures.

     Exclusion Criteria:

A patient who meets any of the following criteria, in either eye, will be excluded from the study:

1. Current or previous myopia treatment with atropine, pirenzepine, or other topical anti-muscarinic
2. Significant central corneal scarring or hydrops
3. Known copper allergy
4. Use of rigid gas permeable lenses, including orthokeratology lenses within 90 days of screening
5. Previous cornea, glaucoma, eyelid, strabismus (exotropia or esotropia) or intraocular surgeries
6. Prior history of ocular disorder (e.g., current or prior history of strabismus (exotropia or esotropia), amblyopia, glaucoma, cataract, retinal detachment or nystagmus, or abnormality of the cornea, lens, iris, ciliary body, or central retina)
7. Myopic degeneration with potential visual acuity worse than Snellen 20/40 (logMAR equivalent 0.3)
8. Intraocular pressure >26 mmHg
9. Medical conditions pre-disposing patient to degenerative myopia or abnormal ocular refractive anatomy (e.g., Stickler Syndrome, Down Syndrome, osteogenesis imperfecta, Ehler's-Danlos Syndrome, Retinopathy of Prematurity)
10. Participation in a clinical trial with use of any investigational drug or treatment within 30 days prior to Visit 1
11. Employees of the study site or their immediate families
12. Pregnancy
13. Hypothyroidism or hyperthyroidism
14. Patient less than 17 Kg weight
15. Planned ophthalmic surgery during the study

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Safety - Change in Best corrected distance visual acuity | Baseline compared to Day 0, Weeks 1, 2 and 4 (+ 5 days)
  Best corrected distance visual acuity in the Study Eye
Phase 1 Safety - Change in Development of corneal scarring | Baseline compared to Day 0, Weeks 1, 2 and 4 (+ 5 days)
  Development of corneal scarring in the study eye
Phase 1 Safety - Change in Patient assessment of comfort | Baseline compared to Day 0, Weeks 1,2 and 4 (+ 5 days)
  Patient assessment of burning, redness, discomfort, irritation in the study eye
Phase 1 Safety - Change in Tyroid enzyme levels | Baseline compared to week 4
  Thyroid enzyme levels
Phase 1 Safety - Change in Copper serum levels | Baseline compared to week 4
  Copper serum levels
Phase 2 Safety - Change in Best corrected distance visual acuity | Weeks 1 and 4 (+ 5 days) and Months 3, 6, 9, and 12 (+ 21 days)
  Best corrected distance visual acuity in the Study Eye
Phase 2 Efficacy - Change/Progression of myopic refractive error | Baseline compared to month 12
  Change/Progression of myopic refractive error (spherical equivalent as determined by cycloplegic refraction) in the Study Eye

SECONDARY OUTCOMES:
Phase 2 Safety - Change in Development of corneal scarring | Weeks 1 and 4 (+ 5 days) and Months 3, 6, 9, and 12 (+ 21 days)
  Development of corneal scarring in the study eye
Phase 2 Safety - Change in Patient assessment of comfort | Weeks 1 and 4 (+ 5 days) and Months 3, 6, 9, and 12 (+ 21 days)
  Patient assessment of burning, redness, discomfort, irritation in the study eye
Phase 2 Efficacy - Change in keratometry | Baseline compared to Weeks 1 and 4 (+ 5 days) and Months 3, 6, 9, 12 (+21 days)
  Measure keratometry in the Study Eye
Phase 2 Efficacy - Change in Axial length | Baseline compared to Weeks 1 and 4 (+ 5 days) and Months 3, 6, 9, 12 (+21 days)
  Axial Length in the Study Eye
Phase 2 Efficacy - Change in Vitreous chamber depth | Baseline compared to Weeks 1 and 4 (+ 5 days) and Months 3, 6, 9, 12 (+21 days)
  Vitreous chamber depth in the Study Eye
Phase 2 Efficacy - Intermediate change/progression of myopic refractive error | Baseline compared to Weeks 1 and 4 (+ 5 days) and Months 3, 6, 9 (+21 days)
  Change/Progression of myopic refractive error (spherical equivalent as determined by cycloplegic refraction) in the Study Eye

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Molokhia, Principal Investigator — iVeena Delivery Systems, Inc.

IPD SHARING:
Plan to Share IPD: No